CLINICAL TRIAL: NCT01884714
Title: New and Innovative Bioanalytical Tools to Assess Lifestyle Recommendations for Managing Type-2 Diabetes
Brief Title: Exploring the Molecular Basis to Healthy Obesity: The Diabetes Risk Assessment Study
Acronym: DRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, David M Mutch, Associate Professor, University of Guelph
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10AP033
Record Dates: First submitted 2013-06-18; First posted 2013-06-24 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Obesity; Type-2 Diabetes; Metabolic Syndrome; Dyslipidemia
Keywords: diabetes; obesity; metabolism; clinical study
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Dyslipidemias; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High fat/high calorie meal (Experimental): All subjects are provided a high calorie (~1300kcal) and high fat (~60g fat) breakfast meal.
  Interventions: Other: High fat/high calorie meal

INTERVENTIONS:
Other: High fat/high calorie meal — All subjects are provided a high calorie (~1300kcal) and high fat (~60g fat) breakfast meal.

SUMMARY:
The purpose of this study is to better understand the genetic and metabolic differences in obese individuals with and without type 2 diabetes. It is expected that this research will help improve our understanding of the variability observed between obese and diabetic individuals.

DETAILED DESCRIPTION:
PURPOSE: Diabetes is one of the fastest growing diseases in Canada; however, lifestyle changes (e.g. changes in diet and physical activity) can prevent or postpone the development of this metabolic disease. The proposed research project hypothesizes that knowledge of the diabetic and obese metabolic phenotype (i.e. the metabotype) has value in predicting these diseases, preventing their downstream complications, and personalizing therapeutic and lifestyle interventions to improve diabetes and obesity management. The overall purpose of this research is to identify biomarkers that uniquely reflect the metabolic perturbations associated with type 2 diabetes and obesity. This information will be invaluable in the design of more personalized interventions to manage these disease states

RATIONALE: Type-2 diabetes is a disease state that affects multiple organs of the biological system, including alterations in adipocyte and muscle insulin signalling, hepatic glucose production, glucose absorption from the gastrointestinal tract, and pancreatic insulin deficiency caused by the loss of β-cell mass and function. Understanding the molecular communication taking place both within and between these tissues is paramount to unravel the metabolic regulatory networks and mechanisms underlying diabetes. Global gene expression profiling (i.e. transcriptomics) and metabolite profiling (i.e. metabolomics) offer powerful approaches to understand the biological processes associated with diabetes and obesity. The analysis of gene expression profiles provides an opportunity to identify early markers of metabolic dysregulation. In contrast, metabolites represent an endpoint of gene and protein function; thus metabolomics is ideally suited for the identification of biomarkers that reflect the biochemical processes underlying a physiological state. By integrating gene expression profiling with metabolite profiling, we will have the opportunity to improve our understanding of the metabolic perturbations related to obesity and/or type-2 diabetes.

OBJECTIVES: The specific goals of this project are to:

1. Recruit a sample of lean, lean/diabetic, obese, and obese/diabetic research participants from the Guelph community.
2. Assess blood glucose and insulin levels in these 4 groups both at baseline and after the consumption of a standardized high fat/high calorie meal.
3. Define the metabotype of these 4 groups by profiling plasma metabolites with mass spectrometry. The current study will examine only blood metabolites.
4. Define subcutaneous adipose tissue gene expression profiles of these 4 groups using microarray technology.

ELIGIBILITY:
Inclusion Criteria:

* Stable body weight (± 2 kg) for at least 3 months.

Exclusion Criteria:

* Evidence of acute or chronic inflammatory disease
* Infectious diseases
* Viral infection
* Cancer
* Alcohol consumption (i.e. more than 2 drinks/day, where 1 drink = 10 g alcohol).

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Measure circulating inflammatory markers and fatty acids associated with obesity and diabetes. | baseline
  Common inflammatory markers (e.g. IL-6, TNFalpha, adiponection) will be measured using either standard ELISA and multiplex bead technology.
  Serum fatty acids will be measured using gas chromatography.

SECONDARY OUTCOMES:
Analyze adipose tissue gene expression in obese and diabetic subjects | baseline
  Gene expression analyzed using microarrays
Measure standard clinical and anthropometric markers associated with obesity and diabetes. | baseline
  Standard clinical parameters (e.g. triglycerides, cholesterol, glucose, insulin, etc) and anthropometric measurements (e.g. body mass index, waist circumference, etc) will be determined.
Examine global serum metabolite profiles associated with obesity and diabetes. | baseline
  Serum metabolites will be measured using gas chromatography coupled with mass spectrometry.
Measure standard clinical and anthropometric parameters in obese and diabetic participants following a standardized meal. | 2 hours after consuming a standardized meal
  All subjects will be provided a standardized meal and after 2 hours standard clinical parameters (e.g. triglycerides, cholesterol, glucose, insulin, etc) will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: David M Mutch, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Human Nutraceutical Research Unit, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perreault M, Zulyniak MA, Badoud F, Stephenson S, Badawi A, Buchholz A, Mutch DM. A distinct fatty acid profile underlies the reduced inflammatory state of metabolically healthy obese individuals. PLoS One. 2014 Feb 10;9(2):e88539. doi: 10.1371/journal.pone.0088539. eCollection 2014. PMID 24520395
- [Result] Badoud F, Lam KP, DiBattista A, Perreault M, Zulyniak MA, Cattrysse B, Stephenson S, Britz-McKibbin P, Mutch DM. Serum and adipose tissue amino acid homeostasis in the metabolically healthy obese. J Proteome Res. 2014 Jul 3;13(7):3455-66. doi: 10.1021/pr500416v. Epub 2014 Jun 23. PMID 24933025
- [Result] Badoud F, Lam KP, Perreault M, Zulyniak MA, Britz-McKibbin P, Mutch DM. Metabolomics Reveals Metabolically Healthy and Unhealthy Obese Individuals Differ in their Response to a Caloric Challenge. PLoS One. 2015 Aug 14;10(8):e0134613. doi: 10.1371/journal.pone.0134613. eCollection 2015. PMID 26274804